CLINICAL TRIAL: NCT06415565
Title: Investigation of the Effectiveness of Thoracic Mobilization Exercise in Fibromyalgia Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uskudar University (Other)
Responsible Party: Principal Investigator, Dr. Öğr. Üyesi Ömer Şevgin, Asst. Prof. Dr., Uskudar University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Uskudar11
Record Dates: First submitted 2024-05-09; First posted 2024-05-16 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: Fibromyalgia
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control (Active Comparator): Conventional physiotherapy practices will be performed.
  Interventions: Other: conventional physiotherapy
- mobilization (Experimental): In addition to conventional physiotherapy applications, thoracic mobilization applications will be performed.
  Interventions: Other: conventional physiotherapy; Other: thoracic mobilization methods

INTERVENTIONS:
Other: conventional physiotherapy — Methods applied as conventional physiotherapy methods are: hotpack, Transcutaneous electrical nerve stimulation and ultrasound.
Other: thoracic mobilization methods — Methods applied as conventional physiotherapy methods: hotpack, Transcutaneous electrical nerve stimulation and ultrasound applications will be applied. Also within the scope of thoracic mobilization: thoracic region extension stretching in the kneeling position, thoracic flexion in the crawling position, halo exercise, thoracic rotation exercises in the crawling position, thoracic rotation in the side lying position. , quadruped extension and rotation exercises will be applied. Patients will be informed that these exercises can also be done as home exercises and they will be asked to practice for 8 weeks.
  Arms: mobilization

SUMMARY:
The aim of this study is to investigate the effects of mobilization exercises applied to the thoracic region on pain, anxiety, depression, disease impact questionnaire, sympathetic and parasympathetic activity in patients diagnosed with fibromyalgia.

DETAILED DESCRIPTION:
The patients included in the study were randomly divided into two as Thoracic Mobilization Group and Control Group and will be included in the treatment programs after the initial evaluations. Patients in both groups will receive a treatment of 11 sessions in total, 5 sessions per week. Participants will be evaluated twice before and after treatment with the Fibromyalgia impact questionnaire, Beck anxiety and Beck depression questionnaires. In addition, the E-motion Faros device will be used to measure heart rate variability. Measurements of heart rate variables will be made before and after the first day of treatment, before and after the 11th session, and on the 45th day.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with fibromyalgia by a specialist physician according to the 2013 American Association of Rheumatology diagnostic criteria
* Being between the ages of 18-45

Exclusion Criteria:

* Those with neurological deficit
* During menopause and postmenstrual period
* Diagnosed with diabetes
* Those with neuropathic disease
* Those with chronic inflammation
* Have immunodeficiency
* Those with cardiac disease
* Patients who are pregnant

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2024-05-15 (Actual); Primary Completion 2024-07-19 (Actual); Study Completion 2024-07-19 (Actual)

PRIMARY OUTCOMES:
Beck Depression Scale | 8 weeks
  The Beck Depression Scale is a 21-item, self-report rating inventory that measures characteristic attitudes and symptoms of depression. The 21 questions in the Beck Depression Scale reflect the symptoms, attitudes and intensity of depression; Items receive a score between zero and three. The total score ranges from 0 to 63. Scores from 0 to 9 indicate no or minimal depression; Scores from 10 to 18 indicate mild to moderate depression; Scores from 19 to 29 indicate moderate to severe depression, and scores from 30 to 63 indicate severe depression.
Beck Anxiety Scale | 8 weeks
  The Beck Anxiety Scale is a self-report questionnaire that measures 21 common somatic and cognitive symptoms of anxiety. Beck Anxiety Scale has 21 questions, each question scored between 0 and 3. The total score to be obtained from the scale varies between 0-63. Beck Anxiety Scale scores are classified as minimal anxiety (0 to 7), mild anxiety (8 to 15), moderate anxiety (16 to 25), and severe anxiety (30 to 63).
Fibromyalgia Impact Survey | 8 weeks
  The Fibromyalgia Impact Questionnaire is an assessment tool developed to measure the condition, progress and outcomes of fibromyalgia patients. It is designed to measure the health status components believed to be most affected in fibromyalgia. Fibromyalgia Impact Questionnaire consists of 10 items. The maximum possible score for each of the 10 items is 10. Therefore the maximum possible score is 100. The average fibromyalgia patient's score is around 50, with severely affected patients often scoring above 70.
Heart rate | 8 weeks
  The E-motion Faros device will be used to measure heart rate variability. E-motion Faros is a 3-electrode device that measures heart rate changes. Two of the electrodes in the device are placed under the patient's right and left clavicle, and the other one is placed just above the lowest left rib. Electrocardiogram measurement takes an average of 5 minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Cansu ÇİFTÇİ, Study Chair — Uskudar University
Locations (1):
- Uskudar Üniversity, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Larsson A, Palstam A, Lofgren M, Ernberg M, Bjersing J, Bileviciute-Ljungar I, Gerdle B, Kosek E, Mannerkorpi K. Resistance exercise improves muscle strength, health status and pain intensity in fibromyalgia--a randomized controlled trial. Arthritis Res Ther. 2015 Jun 18;17(1):161. doi: 10.1186/s13075-015-0679-1. PMID 26084281
- [Background] Bronfort G, Haas M, Evans R, Leininger B, Triano J. Effectiveness of manual therapies: the UK evidence report. Chiropr Osteopat. 2010 Feb 25;18:3. doi: 10.1186/1746-1340-18-3. PMID 20184717
- [Background] Hoogvliet P, Randsdorp MS, Dingemanse R, Koes BW, Huisstede BM. Does effectiveness of exercise therapy and mobilisation techniques offer guidance for the treatment of lateral and medial epicondylitis? A systematic review. Br J Sports Med. 2013 Nov;47(17):1112-9. doi: 10.1136/bjsports-2012-091990. Epub 2013 May 24. PMID 23709519
- [Background] Assumpcao A, Matsutani LA, Yuan SL, Santo AS, Sauer J, Mango P, Marques AP. Muscle stretching exercises and resistance training in fibromyalgia: which is better? A three-arm randomized controlled trial. Eur J Phys Rehabil Med. 2018 Oct;54(5):663-670. doi: 10.23736/S1973-9087.17.04876-6. Epub 2017 Nov 29. PMID 29185675
- [Background] Reis MS, Durigan JL, Arena R, Rossi BR, Mendes RG, Borghi-Silva A. Effects of posteroanterior thoracic mobilization on heart rate variability and pain in women with fibromyalgia. Rehabil Res Pract. 2014;2014:898763. doi: 10.1155/2014/898763. Epub 2014 May 29. PMID 24991436